CLINICAL TRIAL: NCT02538029
Title: The Effects of Dual Task Training on Motor and Non-Motor Function in Individuals With Parkinson's Disease
Brief Title: The Effects of Dual Task Training in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Davis Phinney Foundation (Other)
Responsible Party: Principal Investigator, Jay Alberts, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1000
Record Dates: First submitted 2015-08-17; First posted 2015-09-02 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-02

CONDITIONS: Parkinson's Disease
Keywords: Dual tasking
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual Task Group (Experimental): This group will complete an exercise intervention that involves performing dual tasking activities (simultaneously performing 2 things at once). This group will exercise 3x/wk for 8 weeks.
  Interventions: Behavioral: Dual Task Group
- Single Task Group (Active Comparator): This group will complete an exercise intervention that involves performing single task activities. The participant will perform motor tasks and cognitive tasks individually. This group will exercise 3x/wk for 8 weeks.
  Interventions: Behavioral: Single Task Group

INTERVENTIONS:
Behavioral: Dual Task Group — Performing motor-motor or motor-cognitive tasks at the same time.
  Arms: Dual Task Group
Behavioral: Single Task Group — Performing motor or cognitive tasks alone.
  Arms: Single Task Group

SUMMARY:
The primary aim of the proposed project is to characterize dual tasking (DT) deficits to improve motor, cognitive, and quality of life outcomes in individuals with Parkinson's disease (PD). Phase 1 of the intervention will involve an in-depth gait analysis on 15 individuals with PD. This gait analysis will utilize the Computer Assisted Rehabilitation Environment (CAREN) system, a virtual reality system with a fully integrated 3-D motion capture system. The purpose of Phase 1 is to generalize characteristics of gait and postural control during specific DT conditions. Phase 2 (N=20) involves the clinical translation of these findings. This phase will involve creating a clinical intervention based on the objective information gathered the CAREN system. The intervention will take place 3x/week for a total of 8 weeks. Interventional groups will include: 1) DT clinical group (N=10) and 2) Single task group (N=10). Outcome measures will be used at the beginning and end of the intervention to assess the feasibility and efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic PD
* Able to provide informed consent
* Ability to ambulate ≥ 300ft with or without an assistive device
* Hoehn and Yahr stage 2-4

Exclusion Criteria:

* Undergone any surgical procedure for the treatment of PD, such as deep brain stimulation
* Those who are considered to be high risk exercisers per American College of Sports Medicine exercise screening questionnaire
* Musculoskeletal injury or neurological injury other than PD that would restrict physical activity
* Inability to follow 2 step commands
* Significant cognitive impairment as designated by ≥ 3 errors on the Short Portable Mental Status Questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Penko AL, Barkley JE, Rosenfeldt AB, Alberts JL. Multimodal Training Reduces Fall Frequency as Physical Activity Increases in Individuals With Parkinson's Disease. J Phys Act Health. 2019 Dec 1;16(12):1085-1091. doi: 10.1123/jpah.2018-0595. Epub 2019 Oct 24. PMID 31648204
- [Derived] Rosenfeldt AB, Penko AL, Streicher MC, Zimmerman NM, Koop MM, Alberts JL. Improvements in temporal and postural aspects of gait vary following single- and multi-modal training in individuals with Parkinson's disease. Parkinsonism Relat Disord. 2019 Jul;64:280-285. doi: 10.1016/j.parkreldis.2019.05.021. Epub 2019 May 14. PMID 31103489
- [Derived] Rosenfeldt AB, Penko AL, Bazyk AS, Streicher MC, Dey T, Alberts JL. The Two Minute Walk Test Overground and on a Self-Paced Treadmill Detects Dual Task Deficits in Individuals With Parkinson's Disease. J Aging Phys Act. 2019 Dec 1;27(4):843-847. doi: 10.1123/japa.2018-0264. PMID 31034314

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Will collect in-depth gait assessments under single and dual task conditions. This is a non-interventional group, with all outcomes collected during a single visit.
- Phase 2: Dual Task: This group will complete an exercise intervention that involves performing dual tasking activities (simultaneously performing 2 things at once). This group will exercise 3x/wk for 8 weeks.
- Phase 2: Single Task: This group will complete an exercise intervention that involves performing single task activities. The participant will perform motor tasks and cognitive tasks individually. This group will exercise 3x/wk for 8 weeks.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2: Dual Task | Phase 2: Single Task
Started | 24 | 10 | 11
Completed | 23 | 10 | 10
Not Completed | 1 | 0 | 1
Not completed — unable to complete cognitive assessments | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two participants (one in Phase 1 and one in Phase 2) were unable to complete the required cognitive assessments, and thus were excluded from all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2: Dual Task | Phase 2: Single Task | Total
Number analyzed (Participants) | 23 | 10 | 10 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.61 (7.00) | 58.90 (8.50) | 64.60 (8.46) | 62.74 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 1 | 18
  Male | 11 | 5 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 23 | 10 | 9 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 23 | 10 | 9 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 10 | 10 | 44
Step Length [Mean (Standard Deviation); unit: meters] — The average distance from heel strike of the less affected leg to heel strike of the more affected leg.
  meters | 0.57 (0.14) | 0.63 (0.15) | 0.54 (0.15) | 0.58 (0.14)
Walking Speed [Mean (Standard Deviation); unit: meters/second] — Average self-selected walking speed without dual tasking.
  meters/second | 1.24 (0.14) | 1.19 (0.34) | 1.00 (0.27) | 1.18 (0.14)

OUTCOME MEASURES:

1. Primary Outcome: Step Length During Gait
Description: The average distance from heel strike of the less affected leg to heel strike of the more affected leg. Higher values indicate a longer step length.
Time Frame: Phase 1: baseline; Phase 2: baseline, end of treatment (8 weeks), and end of treatment +4 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Phase 1 | Phase 2: Dual Task | Phase 2: Single Task
Number analyzed (Participants) | 23 | 10 | 10
meters
  Baseline | 0.57 (0.14) | 0.63 (0.15) | 0.54 (0.15)
  End of Treatment: number analyzed (Participants) | 0 | 10 | 10
  End of Treatment |  | 0.72 (0.12) | 0.66 (0.17)
  End of Treatment+4 weeks: number analyzed (Participants) | 0 | 10 | 10
  End of Treatment+4 weeks |  | 0.71 (0.12) | 0.67 (0.16)

2. Primary Outcome: Walking Speed During Gait
Description: Average self-selected walking speed without dual tasking.
Time Frame: Phase 1: baseline; Phase 2: baseline, end of treatment (8 weeks), and end of treatment +4 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Phase 1 | Phase 2: Dual Task | Phase 2: Single Task
Number analyzed (Participants) | 23 | 10 | 10
meters/second
  Baseline | 1.24 (0.21) | 1.19 (0.34) | 1.00 (0.27)
  End of Treatment: number analyzed (Participants) | 0 | 10 | 10
  End of Treatment |  | 1.41 (0.30) | 1.25 (0.35)
  End of Treatment+4 weeks: number analyzed (Participants) | 0 | 10 | 10
  End of Treatment+4 weeks |  | 1.39 (0.30) | 1.29 (0.37)

3. Secondary Outcome: 2 Minute Walk Test
Description: A functional endurance assessment, reporting total distance traveled over a 2 minute period. Higher values indicate better functional endurance.
Time Frame: Phase 1: baseline; Phase 2: baseline, end of treatment (8 weeks), and end of treatment +4 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Phase 1 | Phase 2: Dual Task | Phase 2: Single Task
Number analyzed (Participants) | 23 | 10 | 10
meters
  Baseline | 158.10 (25.98) | 135.28 (21.33) | 134.94 (35.19)
  End of Treatment: number analyzed (Participants) | 0 | 10 | 10
  End of Treatment |  | 147.53 (22.30) | 140.15 (33.18)
  End of Treatment +4 weeks: number analyzed (Participants) | 0 | 10 | 10
  End of Treatment +4 weeks |  | 143.77 (20.35) | 139.27 (31.79)

4. Secondary Outcome: Quality of Life in Neurological Disorders Questionnaire
Description: Quality of life questionnaire. Reported here is T-Score for the Lower Extremity domain. A T-score of 50 is the mean of the reference population, with higher scores indicating a better outcome.
Time Frame: Phase 2: baseline, end of treatment (8 weeks), and end of treatment +4 weeks
Population: One participant in Phase 2 was unable to complete the required cognitive assessments, and thus was excluded from all analyses. One participant did not complete this assessment at EOT+4.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Dual Task | Phase 2: Single Task
Number analyzed (Participants) | 10 | 10
T-score
  Baseline | 43.84 (5.85) | 44.84 (7.69)
  End of Treatment | 45.76 (5.95) | 44.17 (8.10)
  End of Treatment +4 weeks: number analyzed (Participants) | 10 | 9
  End of Treatment +4 weeks | 46.14 (5.96) | 45.85 (7.99)

5. Secondary Outcome: Activities-specific Balance Confidence Scale
Description: Balance questionnaire. Scores range from 0-100, with higher scores indicating greater balance confidence.
Time Frame: Phase 2: baseline, end of treatment (8 weeks), and end of treatment +4 weeks
Population: One participant in Phase 2 was unable to complete the required cognitive assessments, and thus was excluded from all analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: Dual Task | Phase 2: Single Task
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 78.44 (19.34) | 75.44 (22.94)
  End of Treatment | 83.69 (16.92) | 76.44 (18.64)
  End of Treatment +4 weeks | 83.81 (11.19) | 79.38 (15.90)

6. Secondary Outcome: Trail Making Test
Description: Cognitive task where the participant connects 25 dots in numerical order. Lower scores indicate better cognitive function. Reported here is total time to complete the task.
Time Frame: Phase 2: baseline, end of treatment (8 weeks), and end of treatment +4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phase 2: Dual Task | Phase 2: Single Task
Number analyzed (Participants) | 10 | 10
seconds
  Baseline | 31.15 (13.99) | 40.72 (28.22)
  End of Treatment | 28.82 (8.07) | 38.44 (20.44)
  End of Treatment +4 weeks: number analyzed (Participants) | 10 | 9
  End of Treatment +4 weeks | 30.18 (11.68) | 41.57 (25.37)

7. Secondary Outcome: Reaction Time
Description: Average time taken to react to a choice of two stimuli. Lower scores indicate better reaction time.
Time Frame: Phase 2: baseline, end of treatment (8 weeks), and end of treatment +4 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Phase 2: Dual Task | Phase 2: Single Task
Number analyzed (Participants) | 10 | 10
milliseconds
  Baseline | 533.50 (83.85) | 513.44 (129.78)
  End of Treatment | 510.24 (70.94) | 535.76 (119.62)
  End of Treatment +4 weeks: number analyzed (Participants) | 10 | 9
  End of Treatment +4 weeks | 532.49 (88.21) | 558.55 (197.19)

ADVERSE EVENTS:
Time Frame: Phase 1: study duration (1 day) Phase 2: study duration (an average of 13 weeks)
Arm/Group | Phase 1 | Phase 2: Dual Task | Phase 2: Single Task
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/24 | 1/10 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=24) | Phase 2: Dual Task (N=10) | Phase 2: Single Task (N=11)
Fall without injury (General disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02538029/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT02538029/SAP_001.pdf